CLINICAL TRIAL: NCT06666673
Title: Effect of Neural Constraints on Movement in Stroke
Acronym: ENCMS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jun Yao, Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU00223059; 2R01HD039343-16 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Neurotransmitters; flexion synergy; brain plasticity; tizanidine; stroke; motor control; spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — tizanidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): One lactose pill will be administered as a control.
  Interventions: Drug: Placebo
- Drug Probe (Active Comparator): 8 mg Tizanidine
  Interventions: Drug: Tizanidine

INTERVENTIONS:
Drug: Tizanidine — Tizanidine (TIZ) (Zanaflex®) is a centrally acting noradrenergic α-2 agonist and a ligand of I3 (non-I1/I2) imidazoline receptors. It is currently indicated for the management of spasticity.
  Other Names: Zanaflex®
  Arms: Drug Probe
Drug: Placebo — Administered as control
  Arms: Placebo

SUMMARY:
This study investigates the effects of Tizanidine on the voluntary movement controls of the arms of participants who have had a stroke and have not had a stroke by measuring medication-induced changes in upper extremity kinematics, pupillometry, and brain activity. Tizanidine is approved by the U.S. Food and Drug Administration. Understanding how different areas of the brain are involved in movement impairments may help rehabilitation efforts and assist in restoring healthy movement in individuals who have had a stroke.

DETAILED DESCRIPTION:
Sixty-four individuals with stroke will be recruited. Efforts will be made to recruit the same participants for each protocol. A REDCap database for this study will be setup to manage every step involved in the protocol.

The experiment uses a two-arm, cross-over, double-blinded, pre-test-post-test, randomized controlled design. After confirming eligibility, all enrolled participants will be scheduled for one anatomic brain MRI data collection and 6 arm/ hand experiments: 2 for each aim, one with TIZ and the other with placebo. All experiments will take place on separate days at least one week apart. During each of the experimental sessions, the participant will complete the protocol both before and 1.5 hours after administration of either TIZ or a placebo. The order of using TIZ or a placebo will be double-blinded and randomized to balance the FMA of the participants who receive the TIZ or placebo during their first session. In Aim 1, individuals will perform various isometric tasks with their paretic upper limb while high-density surface electromyography is used to estimate the behavior of their motor units. In Aim 2, individuals will perform isometric shoulder abduction with their cortical activity estimated with electroencephalography and their muscle activity recorded with electromyography. In Aim 3, individuals will be placed in a novel robotic device and asked to produce various shoulder abduction torques while either being perturbed by the device to elicit stretch reflexes or asked to perform reaching and hand-opening tasks. For all aims, joint torque and surface electromyographic data will be obtained from each participant before and 1.5 hours after administration of placebo or Tizanidine. Additionally, electroencephalographic data will be obtained during the second aim and joint kinematics will be obtained in the third aim. In all aims, participants will be seated in a Biodex chair (System 3 ProTM; Shirley, New York, USA) with their paretic limb interfaced to a novel haptic device (NACT-3D, Plaisier et. al., 2023) to measure and manipulate the forces/torques experienced by the participant. Throughout each session, straps will be placed across the chest and waist to prevent unwanted movement. The total time from enrollment to completion of participants is expected to be 8-12 weeks, during which participants will be instructed to keep performing routine daily activities.

AE and SAE reporting Adverse event (AE) report form has been implemented in the RedCap database, which can be used at any time. The investigators will report all AEs to the Northwestern Institutional Review Board (IRB) per established policies and requirements. The investigators will create AE reports every six months to review for trends and troubleshoot any issues that arise and require study protocol revision. If any AEs are reported that require follow-up medical care, the investigators will immediately refer the participant back to his/her physician team.

Serious adverse events (SAEs) that are unanticipated, serious, and possibility related to the study intervention will be reported to the Independent Monitor(s), IRB, and National Institute of Child Health and Human Development (NICHD) in accordance with requirements. Unexpected fatal or life-threatening AEs related to the intervention will be reported to the Northwestern IRB in accordance with IRB requirements within 24 hours, and to the NICHD program Officer with 7 days. Other serious and unexpected AEs related to the intervention will also be reported to the Northwestern IRB in accordance with IRB requirements within 24 hours, and to the NICHD program Official within 15 days. Anticipated or unrelated SAEs will be handled in a less urgent manner but will be reported to the PIs, IRB, NICHD, and other oversight organizations in accordance with their requirements. In the annual AE summary, the PIs Report will state that they have reviewed all AE reports.

ELIGIBILITY:
Inclusion Criteria:

* History of unilateral supratentorial ischemic stroke that occurred at least six months prior to enrollment
* Age between 18-80
* Paresis confined to one side, with substantial motor impairment of the upper limb and some residual voluntary movement (Upper Extremity Fugl-Meyer Assessment in the range of 15-45/66, Chedoke McMaster Stroke Assessment Hand section <=4)
* Ability to communicate, understand, and provide informed consent
* Ability to elevate their limb against gravity up to at least 75 degrees of shoulder flexion and to generate active elbow extension
* MRI compatible
* Intact skin on the hemiparetic arm
* Ability to sit for three hours.

Exclusion Criteria:

* Motor or sensory impairment in the non-affected limb (FMA<66, filament >3.6)
* Any brainstem and/or cerebellar lesion
* untreated cardiovascular disease
* History of neurologic disorder other than stroke that affects the arms
* Any acute or chronic painful condition in the upper extremities or spine, indicated by a score ≥5 on a 10-point visual analog scale
* Current use of a pacemaker
* History of seizure
* Chemo denervation: botulinum toxin injection to any portion of the paretic upper extremity within the last 6 months, or phenol/alcohol injections <12 months before participation
* Flexion contractures larger than 30 degrees in the elbow, wrist, metacarpophalangeal joints (MCP) and interphalangeal joints (IP) after stretching for 15 minutes
* Current participation in any experimental rehabilitation or drug studies
* Individuals with any known contraindications to Tizanidine or currently taking Tizanidine; - concurrent use of medications known to suppress central nervous system activity
* pregnant women or women who are nursing.

Additionally, each participant will be asked to provide a list of their current medications and a medical screening questionnaire will be sent to their primary physician. Each participant's list of medications will be reviewed for possible interactions with the study drugs and, at the study physician's advice, will be excluded from the study or asked to withhold medications when applicable. A full list of potential drug interactions can be seen in "Medication Interactions", but concisely includes the following: medications with dopaminergic, serotonergic, or noradrenergic actions; central nervous system (CNS) depressants; antihypertensive/ antiarrhythmic agents; and hormonal medications/contraceptives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Brace Height | Before and 1.5 hours after administration of TIZ
  Brace height quantifies the amplification in motor unit discharge rate generated by PICs. Brace height is sensitive to the level of neuromodulatory drive received by motoneurons.
Cortico-muscular-coherence in beta band | Before and 1.5 hours after administration of TIZ
  Cortico-muscular coherence (CMC) is a commonly used method to measure the synchronized activity between cortex and muscles. Specifically, betaband CMC has been reported to be linked to the use of corticospinal tract.
Difference in reaching distance under shoulder abduction load | Before and 1.5 hours after administration of TIZ
  The difference in reaching distance under shoulder abduction (SABD) load measures the strength of flexion synergy.
Reflexive electromyograph activity prior to movement | Before and 1.5 hours after administration of TIZ
  Reflexive electromyograph (EMG) activity will be calculated as the difference between perturbation-induced EMG amplitude and baseline EMG, averaged during three-time windows 1) before the perturbation -100- 0 ms pre-perturbation; 2) 25 - 75 ms (shortlatency stretch reflex) and 2) 75 - 125 ms (long latency stretch reflex) after the perturbation onset. Perturbations occur at rest before the onset of a regular ballistic reaching trial. EMG is then normalized by the maximal EMG of the corresponding muscle.

SECONDARY OUTCOMES:
Delta-F | Before and 1.5 hours after administration of TIZ
  Delta-F quantifies hysteresis (i.e., prolongation, or persistence) in motor unit firing induced by persistent inward currents (PICs). Delta-F is less selective to the level of neuromodulatory drive, but also accounts for inhibitory synaptic inputs to motoneurons.
Cortico-muscular-coherence in alpha band | Before and 1.5 hours after administration of TIZ
  Alpha-band cortico-muscular-coherence (CMC) has been reported to be linked to the use of cortico-reticulospinal tract. A decreased use of cortico-reticulospinal tract will indirectly reflect an increased use of corticospinal tract, when the require motor task is still performed successfully.
Cortical Laterality Index (LI) | Before and 1.5 hours after administration of TIZ
  LI measures the relatively higher (close to 1) or lower (close to -1) cortical activity between the lesioned vs non-lesioned motor cortices. An increase in LI indicates a shift of cortical activity towards the lesioned motor cortices, and thus reflecting an increased use of corticospinal tract. Minimum value is -1 and maximum value is 1. Higher scores indicate increased use of corticospinal tract.
Difference in Hand hexagon area under SABD load | Before and 1.5 hours after administration of TIZ
  Hand hexagon area (HHA), i.e. the polygon created by connecting the five fingers of the hand with the base of the palm together in a plane, measures hand opening ability. The difference in HHA under SABD load also measures the strength of flexion synergy, but more distally. The investigators hypothesize that the difference under load will become less following tizanidine administration.
Reflexive EMG activity during movement | Before and 1.5 hours after administration of TIZ
  The investigators will calculate the reflexive EMG activity as in Hypothesis 3.2, but with the perturbation occurring during the onset of a ballistic reach.

CONTACTS AND LOCATIONS:
Overall Officials: Julius Dewald, DPT, PhD, Principal Investigator — Northwestern University; Jun Yao, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Dept. of PTHMS 645 N Michigan Ave, Suite 1100, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT06666673/ICF_000.pdf